CLINICAL TRIAL: NCT04759456
Title: Obstructive Sleep Apnea and Comprehensive Remotely-supervised Rehabilitation Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Jakub Hnatiak, MSc., MSc., Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIG 2/20
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Remotely-supervised rehabilitation program; Apnea-Hypopnea Index; Telemonitoring; Telecoaching; Telerehabilitation; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants will undergo 12-week comprehensive remotely-supervised rehabilitation program along with individually titrated CPAP therapy.
  Interventions: Other: Remotely-supervised rehabilitation program
- Control group (No Intervention): Participants will undergo individually titrated CPAP therapy.

INTERVENTIONS:
Other: Remotely-supervised rehabilitation program — Include nutrition, health-related lifestyle and behavioral changes recommendations, and at least 5 times a week 30 minutes of moderate-intensity aerobic training, 10 minutes of inspiratory and expiratory muscle training with breathing device and 10 minutes of oropharyngeal exercise along with individually titrated CPAP therapy
  Arms: Intervention group

SUMMARY:
The purpose of this study is to investigate the feasibility and effect of a 12-week remotely-supervised rehabilitation program in male patients between 25-65 years old with newly diagnosed obstructive sleep apnea with Apnea-Hypopnea Index greater than 15 episodes per hour indicated to CPAP therapy.

DETAILED DESCRIPTION:
The intervention group will undergo comprehensive remotely-supervised rehabilitaiton program in home conditions with teleconsultation (contains telecoaching, telemonitoring) via regular phone calls and e-mails at least 2 times a week. The intervention will include nutrition, health-related lifestyle and behavioral changes recommendations, and at least 5 times a week 30 minutes of moderate-intensity aerobic training, 10 minutes of inspiratory and expiratory muscle training with breathing device and 10 minutes of oropharyngeal exercise along with individually titrated CPAP therapy.

The control group will undergo individually titrated CPAP therapy only. The participants in both groups will go through the following assessments before and after this study: polysomnography, spirometry, anthropometry and body composition examination, laboratory values examination, quality of life questionnaires, Epworth sleepiness scale, 6-min walking test.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* newly diagnosed obstructive sleep apnea
* Apnea-Hypopnea Index greater than 15 episodes/hour
* indicated for CPAP therapy

Exclusion Criteria:

* severe pulmonary hypertension
* severe heart valve disease
* COPD III or IV
* central sleep apnea
* chronic corticosteroid therapy
* long-term oxygen therapy
* heart failure
* left ventricular ejection fraction lower than 40 %
* NYHA III or IV
* cerebrovascular disease
* psychiatric disease
* another type of obstructive sleep apnea treatment
* acute coronary syndrome in anamnesis

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Apnea-Hypopnea Index at Week 12 | Baseline and Week 12
  Measure will be taken from Polysomnography. Index shows number of apneic or hypopneic periods with duration at least 5 seconds in one hour. Higher Index means worse outcome.
Change from Baseline in Epworth Sleepiness Scale Score at Week 12 | Baseline and Week 12
  ESS Score is validated, self-reported instrument of patient's perception of obstructive sleep apnea. Possible scores range is from 0 to 24 points. Higher score means worse outcome.
Change from Baseline in SF-36 Questionnaire Score at Week 12 | Baseline and Week 12
  SF-36 Score is validated, self-reported instrument of patient's perception of health state and quality of life. Possible scores range is from 0 to 100 points. Higher score means better outcome.
Changes from Baseline in Body composition at Week 12 | Baseline and Week 12
  Measure will be taken from InBody 370.
Change from Baseline in 6 Minutes Walking Test at Week 12 | Baseline and Week 12
  6MWT will be evaluated on flat 30 metres long track marked with two cones. Longer distance means better outcome.
Change from Baseline in Maximal Inspiratory Pressure at Week 12 | Baseline and Week 12
  Participants will make 3-5 attempts with 1 minute pause between them. Noted will be the highest score. Higher score means better outcome.
Change from Baseline in Maximal Expiratory Pressure at Week 12 | Baseline and Week 12
  Participants will make 3-5 attempts with 1 minute pause between them. Noted will be the highest score. Higher score means better outcome.

SECONDARY OUTCOMES:
Change from Baseline in Oxygen Desaturation Index at Week 12 | Baseline and Week 12
  Measure will be taken from Polysomnography. ODI means number of times per hour of sleep that the blood's oxygen level drop by a certain degree from baseline.
Change from Baseline in Neck/Waist/Hip circumferences at Week 12 | Baseline and Week 12
  All circumferences will be measured by tape measure.
Change from Baseline in Body Mass Index at Week 12 | Baseline and Week 12
  BMI will be calculated of participant's current weight and height.
Change from Baseline in Forced Vital Capacity at Week 12 | Baseline and Week 12
  Measure will be taken from Spirometry.
Change from Baseline in Forced Expiratory Volume in 1 Second at Week 12 | Baseline and Week 12
  Measure will be taken from Spirometry.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hnatiak J, Zikmund Galkova L, Winnige P, Batalik L, Dosbaba F, Ludka O, Krejci J. Obstructive Sleep Apnea and a Comprehensive Remotely Supervised Rehabilitation Program: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Sep 18;12:e47460. doi: 10.2196/47460. PMID 37721786